CLINICAL TRIAL: NCT02579122
Title: REVIparin-BRIDging-in a General Practice Setting in GErmany (REVIBRIDGE). Non-interventional Study to Evaluate Reviparin for Prevention of Thrombosis and Thromboembolism in General and Orthopedic Surgery (Here: for Perioperative Bridging of Oral Anticoagulation in Interventional Procedures) in General Practices
Brief Title: REVIparin-BRIDging-in a General Practice Setting in GErmany
Acronym: REVIBRIDGE
Status: Terminated | Type: Observational
Why Stopped: Poor recruitment
Sponsor: Mylan Inc. (Industry)
Collaborators: Winicker Norimed GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: DE_2015_REVI_PMOS
Record Dates: First submitted 2015-09-29; First posted 2015-10-19 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2016-08

CONDITIONS: Thromboembolism
Keywords: Reviparin; Bridging; Phenprocoumon
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In view of the fact that little is known about the pre- and post-interventional coagulation management of phenprocoumon patients with reviparin at general practices in Germany, an observational study is being initiated to evaluate the effectiveness and tolerability of reviparin in the area of outpatient, general practice-based care in the context of bridging therapy. Patients for whom bridging therapy with low-molecular weight heparin (LMWH) was specified and for whom the LMWH reviparin was chosen for this purpose shall be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Requiring prophylaxis/bridging treatment with reviparin, e.g. for the prevention of venous thromboembolism in general and orthopaedic surgery, due to the decision of the treating physician

Exclusion Criteria:

* Hypersensitivity to reviparin or one of the excipients of Clivarin® or other low-molecular-weight heparin preparations and/or heparin, e.g. confirmed or suspected immune-mediated heparin-induced thrombocytopenia (type 2)
* Severe renal impairment (creatinine clearance < 30 ml/min)
* Bleeding: like other anticoagulants, reviparin should not be used in conditions associated with an increased risk of bleeding, e.g. acute bleeding, haemorrhagic diathesis, coagulation factor deficiencies, severe thrombocytopenia, untreated arterial hypertension, bacterial endocarditis and subacute endocarditis, acute-onset gastrointestinal ulcers or haemorrhages, brain haemorrhage, spinal or ear or eye surgery, intraocular bleeding or corresponding injuries within the past 6 months
* Severe hepatic or pancreatic impairment
* Children
* Patients with a body weight < 45kg
* Life expectancy of less than 3 months
* Pregnant women (due to the generally very long duration of treatment with LMWH in female patients who are already on anticoagulation therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients under oral anticoagulation with phenprocoumon in general practices
Sampling Method: Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2015-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Patients without thromboembolic or bleeding complications in relation to Reviparin dosage | 15 months
  Documentation of the effect and the dosage of reviparin for the prevention of thromboembolic events in patients on oral anticoagulation (OAC) with phenprocoumon who need to undergo an elective surgical procedure or invasive investigation (target International Normalized Ratio (INR) between 2 and 3) and therefore receive bridging anticoagulation.

SECONDARY OUTCOMES:
Documentation of the bridging regimen with reviparin used in Germany. | 15 months
  mean reviparin dose regimen measured in IU anti-Xa/ per day along with preoperative phenprocoumon withdrawal and postoperative re-onset over the related time course

CONTACTS AND LOCATIONS:
Overall Officials: Alisia Sachse, MD, Study Director — Mylan
Locations (11):
- Germany (11):
  - Research Facility 52, Berlin
  - Research facility 49, Berlin
  - Research facility 136, Essen
  - Research facility 139, Gladbeck
  - Research Facility 163, Herne
  - Research facility 123, Krefeld
  - Research Facility 82, Landsberg
  - Research facility 84, Leipzig
  - Research facility 70, Nossen
  - Research facility 119, Wachtendonk
  - Research facility 125, Wachtendonk